CLINICAL TRIAL: NCT03254628
Title: Saving Lives at Birth in Uganda: Building and Sustaining Capacity of Frontline Health Workers - A Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AID-OAA-A-13-00012
Record Dates: First submitted 2017-07-20; First posted 2017-08-18 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Postpartum Hemorrhage; Neonatal Asphyxia
MeSH Terms: conditions — Postpartum Hemorrhage; Asphyxia Neonatorum | interventions — Oxytocin; Misoprostol; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full - Train/oxy&miso/ B&M/Mentor/Phone (Experimental): Helping Mothers Survive- Bleeding After Birth training and Helping Babies Breathe training done at the facility, simulator present in each facility, oxytocin and misoprostol backfill, newborn bag and mask, designation of Clinical Mentor in each facility to support deliberate practice, phone-based support from district trainer for Clinical Mentor.
  Interventions: Other: Helping Mothers Survive - Bleeding After Birth training; Other: Helping Babies Breathe; Behavioral: Mentor; Behavioral: Phone; Drug: oxytocin and misoprostol; Device: Newborn bag and mask
- Partial - Train/oxy & miso/ B&M/Mentor (Experimental): Helping Mothers Survive - Bleeding After Birth training and Helping Babies Breathe training done at the facility, simulator present in each facility, oxytocin and misoprostol backfill, newborn bag and mask, designation of clinical mentor in each facility to support deliberate practice.
  Interventions: Other: Helping Mothers Survive - Bleeding After Birth training; Other: Helping Babies Breathe; Behavioral: Mentor; Drug: oxytocin and misoprostol; Device: Newborn bag and mask
- Comparison - Train/oxy & miso/ B&M (Active Comparator): Helping Mothers Survive - Bleeding After Birth training and Helping Babies Breathe training done at the facility, simulator present in each facility, oxytocin and misoprostol backfill, newborn bag and mask,.
  Interventions: Other: Helping Mothers Survive - Bleeding After Birth training; Other: Helping Babies Breathe; Drug: oxytocin and misoprostol; Device: Newborn bag and mask

INTERVENTIONS:
Other: Helping Mothers Survive - Bleeding After Birth training — One-day training in postpartum hemorrhage prevention and treatment; this includes instruction to provide oxytocin within one minute of birth to prevent postpartum hemorrhage.
  Other Names: HMS BAB
Other: Helping Babies Breathe — One-day training in neonatal asphyxia management; this includes routine care for the newborn, such as drying and stimulation immediately after birth, and resuscitation of asphyxiated newborns using a bag & mask device.
  Other Names: HBB
Behavioral: Mentor — A birth attendant in the facility is designated as a clinical mentor and encouraged to lead simulator-based practice sessions in the facility after training day.
  Other Names: CM
  Arms: Full - Train/oxy&miso/ B&M/Mentor/Phone; Partial - Train/oxy & miso/ B&M/Mentor
Behavioral: Phone — District trainers telephone clinical mentors and encourage them to lead practice sessions.
  Arms: Full - Train/oxy&miso/ B&M/Mentor/Phone
Drug: oxytocin and misoprostol — This study did not provide uterotonic drugs except in the case of stock out where locally purchased oxytocin and misoprostol were provided only as back up.
  Other Names: oxy&miso
Device: Newborn bag and mask — All facilities were supplied with at least 1 bag and mask for newborn resuscitation. This bag and mask was used for training, practice, and clinical care
  Other Names: B&M

SUMMARY:
The study aims are to evaluate the impact of supportive follow-up strategies for a novel twinned training and capacity-sustaining program among frontline health workers (providers) attending facility-based births in remote and district level health facilities in Uganda. The program is designed to improve provider competencies, provider performance and health outcomes among women giving birth and newborns.

DETAILED DESCRIPTION:
This study will take place in Uganda at Health Centers (level II, III and IV) and District Hospitals, to reach 'frontline' health providers who attend births. This study will take place in districts meeting study criteria in two regions to demonstrate ability to implement in different geographic settings and potential for scale up. It is a quasi-experimental design with three study arms/groups that receive different levels or intensities and modalities of the program intervention.

Briefly, the same simulator-based training will be provided in all three study arms. After the training, a simulator will be left in the health facility, and providers will be encouraged to practice with it regularly. In two of the study arms, specific health workers will be recruited to support the intervention by encouraging their colleagues to practice with the simulator. In one study arm, the practice will be further reinforced through mobile phone-based support. Following is a more detailed description of each of the three components.

Component 1 (Training): Training is composed of two separate training interventions. First, in each study facility, Ugandan master trainers (district trainers) will conduct a single day, simulator-driven training on PPH prevention and treatment; all providers who attend births will be invited to participate. Eight weeks later, in each facility, the same trainers will conduct a one-day, simulator-driven training for prevention and management of asphyxia in the newborn. After each one-day training, simulators will be left at the facility for practice with a corresponding practice schedule.

Component 2 (Peer-led Practice Sessions): On the day the first training (for PPH), 2 birth attendants at the facility will be selected to serve as clinical mentors (CM). The CMs will be trained to encourage their coworkers to participate in 15-minute practice sessions each week for 8 weeks, in which they will use the simulators to practice the skills learned in the one-day training. After the newborn asphyxia training occurs, these same CMs will be trained to support a similar practice schedule for the following 12 weeks - 8 weeks for newborn asphyxia practice and 4 weeks for combined PPH and asphyxia skills practice.

Component 3 (Mobile phone-based support): CMs will be connected to the district trainer via mobile phone for weekly phone calls during the practice periods to provide reminders and support for practice.

ELIGIBILITY:
Inclusion Criteria:

* For Providers: Health providers who attend births in participating health facility and consent to be assessed at the time of enrollment and at several points in time over two years.
* For Clinical mentors: being an experienced skilled birth attendant and likely to remain at the facility during the study period

For Women in Labor and Delivery and Newborns: Women in any stage of labor in participating facility who consent to observation of their delivery and care of their newborn (or consent from the next of kin if the woman is incapacitated and not able to provide consent)

Facility In-charges and Stakeholders: Facility in-charges at sampled health facilities; stakeholders identified by Jhpiego senior managers as being influential in maternal and newborn health policy decisions in Uganda.

Exclusion Criteria:

* Providers: has <1 year of experience, and has plans to be transferred to another facility or leave the facility soon
* Other types of participants: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3440 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in differences: change in use of oxytocin for prevention of postpartum hemorrhage | Baseline, Midline (6 months), Endline (12 months)
  The change in the percentage of women who received oxytocin in correct dose immediately after vaginal birth in three study arms, as assessed by direct clinical observation, using a standardized checklist.

SECONDARY OUTCOMES:
Change in provider performance on simulator-based assessments | Pre-test (before training)- post-test (immediately after training) - midline (6 months)
  The proportion of providers that obtain a passing score on the assessments, based on assessments done by clinical trainers.
Difference in differences: change in care of the mother composite score | Baseline (before training), Midline (6 months), Endline (12 months)
  A composite variable of care provided to laboring mothers, based on direct clinical observation using a standardized checklist.
Difference in differences: change care of the newborn composite score | Baseline (before training), Midline (6 months), Endline (12 months)
  A composite variable of care provided to laboring mothers, based on direct clinical observation using a standardized checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Cherrie Evans, DrPH, Principal Investigator — Jhpiego

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Williams E, Bazant ES, Holcombe S, Atukunda I, Namugerwa RI, Britt K, Evans C. "Practice so that the skill does not disappear": mixed methods evaluation of simulator-based learning for midwives in Uganda. Hum Resour Health. 2019 Mar 29;17(1):24. doi: 10.1186/s12960-019-0350-z. PMID 30925890
- [Derived] Evans CL, Bazant E, Atukunda I, Williams E, Niermeyer S, Hiner C, Zahn R, Namugerwa R, Mbonye A, Mohan D. Peer-assisted learning after onsite, low-dose, high-frequency training and practice on simulators to prevent and treat postpartum hemorrhage and neonatal asphyxia: A pragmatic trial in 12 districts in Uganda. PLoS One. 2018 Dec 17;13(12):e0207909. doi: 10.1371/journal.pone.0207909. eCollection 2018. PMID 30557350

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-12-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03254628/Prot_SAP_000.pdf
  • Informed Consent Form (2015-02-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03254628/ICF_001.pdf